CLINICAL TRIAL: NCT06386588
Title: The Effects of Auditory Stimulation During Sleep on Offline Learning and Thalamocortical-hippocampal Connectivity in Schizophrenia
Brief Title: The Effects of Auditory Stimulation During Sleep on Brain Networks in Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dara S. Manoach, PhD, Professor, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2024P000610
Record Dates: First submitted 2024-03-28; First posted 2024-04-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia
Keywords: Hippocampus; Neuromodulation; Sleep spindles; Thalamocortical circuits; Auditory stimulation; Magnetic resonance imaging; Sleep; Memory
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schizophrenia (Experimental): Adult outpatients with a diagnosis of schizophrenia.
  Interventions: Other: Closed loop auditory stimulation during sleep
- Healthy Controls (Active Comparator): Adult participants screened to exclude a personal history of mental illness, family history of schizophrenia spectrum disorder, and psychoactive medication use.
  Interventions: Other: Closed loop auditory stimulation during sleep

INTERVENTIONS:
Other: Closed loop auditory stimulation during sleep — Short bursts of pink noise delivered at precise times during overnight sleep at home.

SUMMARY:
In this research study the investigators will use sleep headbands to measure brain rhythms and to improve their coordination across brain regions. The headbands will be worn at home for multiple nights. On some nights the headbands will play soft sounds at specific times during sleep. The investigators are interested in learning whether this timed auditory stimulation may be a strategy to improve the coordination of sleep rhythms across brain regions, improve network communication, and as a result, improve memory. The investigators will study 30 adults aged 18-45 with schizophrenia and 30 demographically matched healthy controls. Participants will first have a daytime MRI scan, during which they will complete a finger tapping motor sequence task (MST), followed by a week of sleep at home with a sleep headband. They will also do the MST at home on two of the nights. On the final day of the study, participants will return for a second MRI scan.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* Fluent in English
* Able to give informed consent

Additional inclusion for Adults with schizophrenia:

* A DSM-V confirmed diagnosis of schizophrenia
* Unmedicated or maintained on a stable dose of APDs

Exclusion Criteria:

* Ferrous metal in the body
* Currently pregnant or breastfeeding
* Motor problems that preclude finger tapping task
* IQ <85
* Other neurological disorders, including seizure disorder
* Significant hearing or vision loss
* Chronic medical conditions that affect sleep
* Unstable chronic medical condition such as asthma, diabetes, cystic fibrosis, or cardiac disease
* Diagnosed sleep disorder, except insomnia
* History of head injury resulting in prolonged loss of consciousness or other neurological sequelae

Additional Exclusion Criteria for Healthy adults:

* History of mental illness
* Current use of psychotropic medications or treatment with medications known to affect sleep or cognition

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in sleep physiology | across 5 nights of sleep with auditory stimulation
  Changes in slow oscillations, sleep spindles, and slow oscillation-spindle coupled events as measured by sleep EEG headband
Changes in functional connectivity of the hippocampus and thalamus | Approximately 1 week between baseline and follow-up scans
  Changes in functional connectivity of the hippocampus and thalamus as measured by resting state functional connectivity MRI
Changes in hippocampal activation during motor sequence task (MST) | Approximately 1 week between baseline and follow-up scans
  Changes in hippocampal activation during the MST as measured by functional MRI
Changes in hippocampal microstructural integrity | Approximately 30 minutes between pre- and post-task diffusion-weighted MRI scans
  Changes in hippocampal microstructural integrity as measured by diffusion-weighted MRI

SECONDARY OUTCOMES:
Greater gains in typing speed over rest breaks during MST training (micro-offline gains) | Approximately 5 days between pre- and post-stimulation MST administrations
  MST training sessions prior to sleep consisting of typing trials separated by rest periods. We will measure typing speed before and after rest breaks.
Sleep dependent memory consolidation (SDMC) | Approximately 5 days between pre- and post-stimulation MST administrations
  Comparison of SDMC between the Baseline MST only and MST with CLASS nights

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No